CLINICAL TRIAL: NCT01710384
Title: Effect of Antenatal Corticosteroids in Late Preterm
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 006111
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Late Preterm
Keywords: late preterm, betamethasone,
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- betamethasoneb, 34-36 weeks, preterm labor (Experimental): betamethasone 12 mg 2 injections will be given 24-hours apart.
  Interventions: Drug: betamethasone
- preterm labor, 34-37 weeks (No Intervention): betamethasone 12 mg 2 injections will be given 24-hours apart.

INTERVENTIONS:
Drug: betamethasone
  Arms: betamethasoneb, 34-36 weeks, preterm labor

SUMMARY:
To test the effect on premature infants of a one-time course of betamethasone administered in weeks 34-36 of gestation.

DETAILED DESCRIPTION:
Protocol version 3, 1/7/2012

Research Goal To test the effect on premature infants of a one-time course of betamethasone administered in weeks 34-36 of gestation.

Inclusion criteria

1. Pregnant woman in weeks 34-36 of gestation who did not receive a betamethasone course to enhance fetal lung maturity during pregnancy
2. Clinical, sonographic or laboratory suspicion of premature labor
3. Singleton or twin pregnancy Exclusion criteria

1. Premature rupture of membranes 2. Fetus with known defects 3. Suspicion of fetal distress 4. Betamethasone administered during pregnancy for any reason Research protocol Study group 100 women in weeks 34-36 of gestation with clinical, sonographic or laboratory suspicion of early labor will be recruited.

Demographic data will be collected, including full medical and obstetrical anamnesis.

After full obstetric analysis, including monitoring, sonographic and lab tests as needed for each case and as determined by department policy, a full course of 2 injections of betamethasone will be given 24-hours apart.

After birth, data will be collected on the delivery, including birth week, method (vaginal, cesarean, forceps, etc.), obstetric complications (abruption of the placenta, Premature rupture of membranes, preeclampsia, etc.). Data on the neonate, including birth weight, 1 and 5 minute Apgar scores, and complications during the first week of life, including hypoglycemia, seizures, intubation or medications will also be collected.

Prospective control group 100 women will be recruited who delivered in the hospital during the study period in weeks 34-37 of pregnancy, who did not receive a course of betamethasone during pregnancy.

Demographic data will be collected, full medical and obstetric anamnesis including current and previous pregnancies.

After birth, data will be collected on the delivery, including birth week, method (vaginal, cesarean, forceps, etc.), obstetric complications (abruption of the placenta, Premature rupture of membranes, preeclampsia, etc.). Data on the neonate, including birth weight, 1 and 5 minute Apgar scores, and complications during the first week of life, including hypoglycemia, seizures, intubation or medications will also be collected.

Data will be collected over a one-year period. Retrospective control group 200 women who delivered from 2009 to 2011, in weeks 34-37 of gestation who did not receive a course of betamethasone during the pregnancy.

Data will be anonymously collected from medical records, including demographics and full medical and obstetric anamnesis.

After birth, data will be collected on the delivery, including birth week, method (vaginal, cesarean, forceps, etc.), obstetric complications (abruption of the placenta, Premature rupture of membranes, preeclampsia, etc.). Data on the neonate, including birth weight, 1 and 5 minute Apgar scores, and complications during the first week of life, including hypoglycemia, seizures, intubation or medications will also be collected.

The pregnancy and neonatal outcomes among the groups of women who received and did not receive betamethasone will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman in weeks 34-36 of gestation who did not receive a betamethasone course to enhance fetal lung maturity during pregnancy 2. Clinical, sonographic or laboratory suspicion of premature labor 3. Singleton or twin pregnancy

-

Exclusion Criteria:

1. Premature rupture of membranes
2. Fetus with known defects
3. Suspicion of fetal distress
4. Betamethasone administered during pregnancy for any reason

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
neonate respiratory distress syndrome | 1 year

SECONDARY OUTCOMES:
1 and 5 minute Apgar scores, and complications during the first week of life, including hypoglycemia, seizures, intubation or medications | 1 week